CLINICAL TRIAL: NCT04919005
Title: Virtual Environment to Aid Cognitive Stimulation of Elderly People With Early Alzheimer's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Associate Professor, University of Mogi das Cruzes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 54290416.9.0000.5497
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy elderly people (Experimental): Twelve healthy elderly people. Each participant underwent a pre-test, the intervention with a Virtual Environment, and a post-test.
  Interventions: Other: Virtual Environment
- Elderly people with Alzheimer's in the initial phase (Experimental): Seven elderly people with Alzheimer's in the initial phase. Each participant underwent a pre-test, the intervention with a Virtual Environment, and a post-test.
  Interventions: Other: Virtual Environment
- Healthy young people (Experimental): Fifteen healthy young people. Each participant underwent a pre-test, the intervention with a Virtual Environment, and a post-test.
  Interventions: Other: Virtual Environment

INTERVENTIONS:
Other: Virtual Environment — The Virtual Environment was called SorrisoTur and consists of 10 mini-games with difficulty levels in a limited number of cities and mini-games distributed in a thematic scenario of the map of Brazil. The virtual environment consists of the cognitive training mini-games within a theme for all screens, mini-games, and information. The interventions with the Virtual Environment were administered in periods of one hour, twice a week, for a month.

SUMMARY:
This research was carried out with the objective of verifying the possibility of intervention through cognitive training protocols to assist in the stimulation of neurons and to delay the degradation resulting from Alzheimer's disease in its initial phase. The specific objective of this research was to develop and validate a virtual environment of games (called SorrisoTur) that allows the intervention of cognitive training.

DETAILED DESCRIPTION:
SorrisoTur encompasses cognitive training concepts and protocols in playful situations, which were coded in the form of 2D mini-games that are run on a computer connected to the Web, and designed to stimulate cognitive domains, such as memory, executive functions, spatial-visual skills, language (expression, comprehension, reading, and writing) and personality/behavior. For the comparison of results, three groups were created; one group of elderly people with Alzheimer's disease at an early stage, one group formed by healthy elderly, and another group with young people and applied Mini-Mental State Examination (MMSE) and Wechsler Intelligence Scale for Adults (WAIS-III) before and after of interventions with the games.

ELIGIBILITY:
Inclusion Criteria:

* People with physical or psychological conditions allow interacting with digital games;
* Elderly over 60 years with mild Alzheimer;
* Seniors over 60 Healthy;
* Healthy Youth;

Exclusion Criteria:

* People without physical or psychological conditions allow interacting with digital games;
* Elderly people over 60 years old who have any type of dementia other than Alzheimer, or moderate or severe Alzheimer;

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Change on Wechsler Intelligence Scale for Adults (WAIS-III) | Baseline and after 4 weeks
  The WAIS-III is an intellectual assessment that aims to analise the measures of the following Factorial Scales and Indexes: Verbal IQ (intelligence quotient), Execution IQ, Total IQ, Verbal Understanding Index, Perceptual Organization Indexes, Operational Memory Indexes and Processing speed index.
Change on Mini Mental State Examination (MMSE) | Baseline and after 4 weeks
  The MMSE is a data collection instrument widely used in cases of dementia, it evaluates temporal and spatial orientation, short-term memory (immediate or attention) and skills of evocation, calculation, praxis, visuospatial, communication and language.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia A Bissaco, PhD, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Terigi Augusto Scardovelli, Mogi das Cruzes, São Paulo, Brazil